CLINICAL TRIAL: NCT04179591
Title: Comparison of the Effects of Foot Exercise Program and Arch Support Insoles on Foot Posture, Plantar Force Distribution, and Balance in Individuals With Flexible Pes Planus
Brief Title: Effects of Exercise and Insole on Foot Posture, Plantar Force Distribution, and Balance in Individuals With Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Müge KIRMIZI, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Müge KIRMIZI
Record Dates: First submitted 2019-11-24; First posted 2019-11-27 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Pes Planus
Keywords: Pes planus; Foot posture; Plantar pressure variables; Balance; Short foot exercises; Tibials posterior strengthening; Intrinsic foot muscles; Custom-made insole; Arch support insole
MeSH Terms: conditions — Flatfoot | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Experimental): Exercises will be performed three times per week for six weeks.
  Interventions: Other: Exercise
- Insole (Experimental): Customized arch support insoles will be worn for six weeks.
  Interventions: Other: Orthesis
- Exercise plus Insole (Experimental): Exercises will be performed three times per week, and customized arch support will be worn for six weeks.
  Interventions: Other: Exercise; Other: Orthesis

INTERVENTIONS:
Other: Exercise — Intrinsic foot muscles and tibialis posterior strengthening exercises
  Arms: Exercise; Exercise plus Insole
Other: Orthesis — Customized arch support insoles
  Arms: Exercise plus Insole; Insole

SUMMARY:
The aim is to compare the effects of intrinsic foot muscles and tibialis posterior strengthening exercise, and customized arch support insoles on foot posture, plantar force distribution, and balance in individuals with flexible pes planus.

DETAILED DESCRIPTION:
The aim is to compare the effects of intrinsic foot muscles and tibialis posterior strengthening exercise, and customized arch support insoles on foot posture, plantar force distribution, and balance in individuals with flexible pes planus. Forty-two individuals with flexible pes planus will be recruited into the study according to the inclusion criteria. Participants will be randomly divided into three groups: (1) Exercise, (2) Insole, (3) Exercise plus Insole. Exercises will be performed three times per week for six weeks, also custom-made insoles will be worn for six weeks. Foot posture will be assessed using the Navicular drop, Valgus index and Foot posture index-6. Plantar force variables will be recorded by the pressure-sensitive mat (HR Mat, Tekscan, USA) mounted in the middle of the 6-meter walkway in three sessions: (1) Upright standing, (2) Walking at different speeds: self-selected slow, normal and fast speeds, (3) Walking just after the heel-rise test for endurance. Balance performance will be assessed by the Balance Master System (NeuroCom® International Inc., USA). The assessments will be made pre/post intervention and at 6-weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. being between 18 and 40 years of age,
2. having Navicular drop test greater than 10 mm,
3. having Foot posture index-6 greater than or equal to 6,
4. having bilateral flexible pes planus.

Exclusion Criteria:

1. a lack of anatomical integrity of the foot,
2. a history of surgery or trauma in the foot region,
3. other musculoskeletal or neurological problems which may affect balance and gait performance.
4. having received any treatment for lower extremity disorders including pes planus within the last 1 year
5. having a body mass index equal to or greater than 30.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Foot posture | Change in foot posture measures from baseline to six weeks and to twelve weeks
  Foot posture will be assessed using the Navicular drop, Valgus index and Foot posture index-6.
Balance | Change in balance scores from baseline to six weeks and to twelve weeks
  Balance performance will be assessed by the Balance Master System (NeuroCom® International Inc., USA).
Plantar force variables | Change in plantar pressure variables from baseline to six weeks and to twelve weeks
  Plantar force variables will be recorded by the pressure-sensitive mat (HR Mat, Tekscan, USA) mounted in the middle of the 6-meter walkway in three sessions: (1) Upright standing, (2) Walking at different speeds: self-selected slow, normal, and fast speeds, (3) Walking just after the heel-rise test for endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Institute of Health Sciences, Izmir, Turkey (Türkiye)